CLINICAL TRIAL: NCT02224638
Title: Evaluation of Wound Management for Sacral Pressure Ulcers With Necrotic Tissue
Brief Title: Wound Management for Sacral Pressure Ulcers With Necrotic Tissue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R14-028
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Pressure Ulcers
Keywords: skin ulcers
MeSH Terms: conditions — Pressure Ulcer; Skin Ulcer | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: A single-center, randomized open-label study with multiple application treatment of necrotic sacral or buttocks pressure ulcers with either TheraHoney HD or SkinTegrity Hydrogel.
Oversight: Data Monitoring Committee: No

ARMS (2):
- TheraHoney HD (Active Comparator): Honey product
  Interventions: Device: TheraHoney HD
- SkinTegrity (Active Comparator): Skin moisturizer
  Interventions: Device: SkinTegrity

INTERVENTIONS:
Device: TheraHoney HD — Honey
  Arms: TheraHoney HD
Device: SkinTegrity — Hydrogel
  Other Names: Hydrogel
  Arms: SkinTegrity

SUMMARY:
Evaluation of a wound care debridement product and a moisturizer on sacral pressure ulcer wounds

DETAILED DESCRIPTION:
Pressure ulcers on the sacral area will be applied with either a wound debridement product or a wound moisturizer product plus a gentle wound dressing to manage wound closure over a 2-3 week period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any age
* Sacral wounds with necrotic tissue

Exclusion Criteria:

* 3rd degree burns
* know hypersensitivity to products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chaiken, RN, Principal Investigator — Swedish Covenant Hospital
Locations (2):
- United States (2):
  - Swedish Covenant Hospital, Chicago, Illinois
  - Harmony Residential Facility, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TheraHoney HD | SkinTegrity
Started | 11 | 10
Completed | 10 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TheraHoney HD | SkinTegrity | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wounds Healed
Description: Percentage of wounds that were complete or partially healed with either treatment measured by change in wound size of sacral pressure ulcer
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: percentage of wounds
Arm/Group | TheraHoney HD | SkinTegrity
Number analyzed (Participants) | 11 | 10
percentage of wounds | 63.1 (38.4) | 6.1 (74.7)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events related to the presence or absence of wound infections and worsening in ulcer staging.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TheraHoney HD | SkinTegrity
Number analyzed (Participants) | 11 | 10
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: wound treatment period of 34 days
Arm/Group | TheraHoney HD | SkinTegrity
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/10
Other Adverse Events (participants affected / at risk) | 1/11 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraHoney HD (N=11) | SkinTegrity (N=10)
Infection/sepsis (Infections and infestations) | 0 (0) | 1 (1)
Ischemic Bowel Surgery (Gastrointestinal disorders) | 1 (1) | 0 (0)
AFIB (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TheraHoney HD (N=11) | SkinTegrity (N=10)
Periwound Maceration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased Wound Size (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No